CLINICAL TRIAL: NCT06050954
Title: GU-216: A Pilot Study of Circulating Tumor DNA Adaptive Risk Maintenance Approach for Bladder Cancer (CARMA)
Brief Title: A Pilot Study of Circulating Tumor DNA Adaptive Risk Maintenance Approach for Bladder Cancer (CARMA)
Acronym: CARMA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in standard of care.
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-1026
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Maintenance Therapy 200mg Pembrolizumab (Other): Participants who have radiographical or ctDNA progression after 3-6 cycles of standard-of-care platinum-based chemotherapy will be offered 200mg Pembrolizumab every six weeks via IV infusion.
  Interventions: Drug: Pembrolizumab (200mg)
- Maintenance Therapy 400mg Pembrolizumab (Other): Participants who have radiographical or ctDNA progression after 3-6 cycles of standard-of-care platinum-based chemotherapy will be offered 400mg Pembrolizumab every six weeks via IV infusion..
  Interventions: Drug: Pembrolizumab (400mg)
- Active Surveillance (Other): Participants who are deemed ctDNA responders (reduction in ctDNA by 50% or more) on post-chemo testing will undergo active surveillance and continued serial ctDNA testing at regular intervals as defined by the study protocol. Patients will also undergo surveillance imaging as defined in the study protocol. At the time of first radiographic or ctDNA progression (to be assessed every 12 weeks in conjunction with radiographic assessment), the patient will be offered treatment with pembrolizumab.
  Interventions: Diagnostic Test: Monitoring

INTERVENTIONS:
Drug: Pembrolizumab (200mg) — 200mg Pembrolizumab every six weeks via IV infusion.
  Arms: Maintenance Therapy 200mg Pembrolizumab
Drug: Pembrolizumab (400mg) — 400mg Pembrolizumab every six weeks via IV infusion.
  Arms: Maintenance Therapy 400mg Pembrolizumab
Diagnostic Test: Monitoring — active surveillance and monitoring via continued serial ctDNA testing and radiographic assessments at regular intervals.
  Arms: Active Surveillance

SUMMARY:
Platinum-based chemotherapy remains the standard of care for advanced/metastatic unresectable bladder cancer. The JAVELIN Bladder 100 and HCRN GU14-182 trials showed that maintenance immune checkpoint inhibition(ICI) for those that achieved disease control could prolong progression-free survival (overall survival benefit in JAVELIN may have been related to the lack of guaranteed crossover at time of progression). Of note, both of these studies showed consistency with regards to the magnitude of the PFS benefit which was ~40% vs ~20% at 6-months with maintenance ICI compared to BSC/placebo. Maintenance avelumab is now category 1 on the NCCN guidelines.

However, some patients prefer prolonged chemotherapy responses and literature supports a treatment break without effecting longevity. The underlying risk resides in the selection of patients with some (currently difficult to diagnose) progressing rapidly. This trial proposes to use ctDNA to stratify chemo-responsive patients to active surveillance (i.e. a ctDNA responder referred to here as "ctDNA-") vs SOC maintenance pembrolizumab (ctDNA+). All patients will be treated with SOC chemotherapy and only patients with an objective (RECIST) response will be stratified.

This is a non-randomized phase 2 study with two arms based on ctDNA

1. Pembrolizumab (ctDNA non-responder) maintenance therapy arm (SOC)
2. Active surveillance arm (ctDNA responders) with serial ctDNA and crossover 1st line chemotherapy is based on physician discretion choice as described in the protocol. Patients with metastatic Urothelial Cancer are enrolled prior to initiation of SOC chemotherapy. Based on ORR (CR + PR), it is estimated that 75 patients will need to enroll onto the protocol to find 25 responders for the two arms.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, unresectable locally advanced or metastatic transitional cell carcinoma of the urothelium.
2. Subjects must be deemed eligible for standard first-line platinum-based chemotherapy for advanced or metastatic urothelial cancer (e.g., as per NCCN guidelines). Eligible regimens include; dose-dense MVAC, gemcitabine + cisplatin and/or gemcitabine + carboplatin. (split-dose dosing of cisplatin for dose-dense MVAC and gemcitabine + cisplatin is allowed)
3. Must have measureable disease per RECIST v1.1.
4. Male or female participants with age ≥ 18 years
5. ECOG performance status 0 or 1.
6. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 6 months after the last dose of study treatment
7. Adequate Bone marrow function:

   1. Absolute neutrophil count (ANC) ≥ 750 /mm3 or ≥0.5 x 109/L
   2. Platelets ≥50,000/mm3 or ≥100 x 109/L
   3. Hemoglobin ≥7.5 g/dL (may have been transfused)
8. Adequate renal function, defined as estimated creatinine clearance ≥ 45 mL/min (calculated using the Cockcroft-Gault formula or measured with 24-hour urine collection)
9. Adequate liver function:

   1. Total serum bilirubin < 1.5 X ULN (Pts with Gilbert's can enroll if conjugated bilirubin is within normal limits)
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 X institutional ULN
10. Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

1. Prior systemic chemotherapy or radiation therapy for advanced or metastatic urothelial carcinoma.
2. Prior immunotherapy with IL-2, IFN-α, or an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA-4 antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
3. Major surgery ≤ 4 weeks or major radiation therapy ≤ 2 weeks prior to enrollment.
4. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided it has not been completed within 48 hours prior to patient enrollment.
5. Participants with known symptomatic central nervous system (CNS) metastases requiring steroids. Participants with previously diagnosed CNS metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to randomization, have discontinued corticosteroid treatment for these metastases for at least 4 weeks, and are neurologically stable
6. Persisting toxicity related to prior therapy NCI CTCAE v5.0 Grade >1; however, sensory neuropathy Grade ≤ 2 is acceptable.
7. On active treatment for any other malignancy, except for adjuvant hormone therapy for localized breast cancer or castration for hormone sensitive prostate cancer.
8. Participation in other studies involving investigational drug(s) within 4 weeks prior to randomization. Observational studies are permitted.
9. History of uncontrolled autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with well-controlled autoimmune disease and mild symptoms on a stable dose of prednisone (≤ 10 mg daily) are allowed on study.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (defined by current oral or intravenous antibiotic therapy), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Patients with prior allogeneic hematologic transplant
12. Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are progression-free by RECIST 1.1 and alive at six months from initiation of active surveillance. | 6 months

SECONDARY OUTCOMES:
Overall survival from initial assignment to active surveillance or maintenance arms defined as time to death (or last known alive) | Up to participant death
Progression-free survival, from initial assignment to maintenance arm defined by RECIST 1.1 or death from any cause. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Miron, Principal Investigator — Fox Chase Cancer Center

IPD SHARING:
Plan to Share IPD: No